CLINICAL TRIAL: NCT03316898
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Determine the Safety, Tolerability, Pharmacokinetics, and Brain Metabolic Response, Using FDG-PET, Following Administration of AGN-242071 Added to Standard-of-Care (Donepezil ± Memantine) in Participants With Mild to Moderate Alzheimer's Disease
Brief Title: A FDG-PET Study of AGN-242071 Added to Standard-of-Care (Donepezil ± Memantine) for the Treatment of Participants With Mild to Moderate Alzheimer's Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision to stop the study.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3142-101-001
Record Dates: First submitted 2017-10-18; First posted 2017-10-20 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil; Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Two placebo capsules once daily for 28 Days. All participants are on a stable dose of 10 mg donepezil and, if receiving memantine, also on a stable dose of memantine as prescribed by the physician as per standard of care.
  Interventions: Drug: Placebo; Drug: Donepezil; Drug: Memantine
- AGN-242071 5 mg (Experimental): One AGN-242071 5 mg capsule plus one placebo capsule once daily for 28 days. All participants are on a stable dose of 10 mg donepezil and, if receiving memantine, also on a stable dose of memantine as prescribed by the physician as per standard of care.
  Interventions: Drug: AGN-242071; Drug: Placebo; Drug: Donepezil; Drug: Memantine
- AGN-242071 15 mg (Experimental): AGN-242071 starting at a dose of one 5 mg capsule plus one placebo capsule once daily for 5 days followed by AGN-242071 15 mg total dose (one 5 mg and one 10 mg capsules) once daily on Days 6 to 28. Dose can be adjusted based on safety and tolerability. All participants are on a stable dose of 10 mg donepezil and, if receiving memantine, also on a stable dose of memantine as prescribed by the physician as per standard of care.
  Interventions: Drug: AGN-242071; Drug: Placebo; Drug: Donepezil; Drug: Memantine
- AGN-242071 25 mg (Experimental): AGN-242071 starting at a dose of one 5 mg capsule plus one placebo capsule once daily for 5 days followed by AGN-24071 15 mg total dose (one 5 mg and one 10 mg capsules) once daily on Days 6 to 10 followed by AGN-242071 25 mg total dose (one 5 mg and one 20 mg capsules) on Days 11 to 28. Dose can be adjusted based on safety and tolerability. All participants are on a stable dose of 10 mg donepezil and, if receiving memantine, also on a stable dose of memantine as prescribed by the physician as per standard of care.
  Interventions: Drug: AGN-242071; Drug: Placebo; Drug: Donepezil; Drug: Memantine

INTERVENTIONS:
Drug: AGN-242071 — AGN-242071 capsules administered once daily to patients receiving donepezil 10 mg with or without memantine as prescribed per standard of care.
  Arms: AGN-242071 15 mg; AGN-242071 25 mg; AGN-242071 5 mg
Drug: Placebo — Placebo capsules once daily to patients receiving donepezil 10 mg with or without memantine as prescribed per standard of care.
Drug: Donepezil — Donepezil 10 mg as prescribed by the physician as per standard of care.
Drug: Memantine — Memantine as prescribed by the physician as per standard of care.

SUMMARY:
This is a study to evaluate the brain metabolic response using Fluorodeoxyglucose Positron Emission Tomography (FDG-PET), safety, tolerability and pharmacokinetics of AGN-242071 in patients with mild to moderate Alzheimer's Disease on a stable dose of 10 mg donepezil with or without memantine standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic evidence of probable Alzheimer's Disease (AD) per the 2011 National Institutes of Aging-Alzheimer's Association (NIA-AA) criteria
* Participants receiving donepezil at a stable dose of 10 mg daily with or without stable dose memantine for at least 6 weeks prior to the screening visit.

Exclusion Criteria:

* Participants with illness apart from AD that could contribute to cognitive dysfunction
* History of clinically significant suicidal ideation within the past 6 months
* Thyroid disease unless the participant is euthyroid and stable on treatment for at least 3 months prior to screening
* Participants with a personal or family history of congenital long QT syndrome or sudden death
* Clinically significant cardiovascular disease in the past 6 months prior to screening
* Participants with signs and symptoms of peripheral vascular disease (PVD)
* A transient ischemic attack or other acute ischemic event affecting the brain, spinal cord, or peripheral circulation in the past 6 months prior to screening
* Any history of cerebrovascular accident or stroke
* Any history of a seizure disorder other than a single febrile seizure
* Pulmonary disease or evidence of clinically significant moderate or severe pulmonary symptoms
* History of cancer within the last 5 years
* Evidence or history of diabetes mellitus Type 1
* Any significant sensory (eg, moderate to severely impaired hearing or severely impaired vision) or hand movement difficulties that would prevent participants from completing the behavioral assessments of the study
* Treatment with cholinesterase inhibitors other than donepezil or other cholinomimetics within 12 weeks of the baseline visit
* Treatment with memantine not in combination with donepezil within 12 weeks of the baseline Visit
* Participants who have been on anticholinergic and/or antimuscarinic treatment including overactive bladder treatments, antihistamines, antipsychotics, and tricyclic antidepressants, within 12 weeks prior to the baseline visit
* Participants who have been on drugs that are strong inhibitors of CYP2D6 or CYP2C9 (eg, quinidine, paroxetine, fluoxetine, terbinafine, bupropion), or that are moderate or strong inhibitors of CYP3A4 (eg, erythromycin, ketoconazole, rifampicin, fluconazole, carbamazepine) within 21 days prior to the baseline visit
* Participants who are taking any moderate or strong inducers of CYP3A4 (eg, carbamazepine, phenytoin, rifampin, modafinil, and herbal preparations containing St. John's wort) or strong inducers of CYP2C9 within 21 days prior to the baseline visit
* Participants who have been on other drugs that could affect cognition (eg, benzodiazepines or gamma-aminobutyric acid A (GABAA) receptor agonists used as anxiolytics, sedative-hypnotics) or over-the-counter (OTC) sleeping aids within 12 weeks prior to the baseline visit
* Participants who have been on hormone replacement therapy, thyroid supplement, vitamin E, or vitamin B12 unless at a stable dose for 4 weeks before the baseline visit
* Use of an active Alzheimer's disease vaccine within 2 years prior to screening or monoclonal antibody for treatment of AD within 1 year prior to screening
* Positive test results for anti-human immunodeficiency virus (anti-HIV) type 1 and 2, hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (anti-HCV) at screening
* Positive test results for urine drug screen for methadone, cocaine, tetrahydrocannabinol, benzodiazepines, tricyclic antidepressants, barbiturates, phencyclidine, amphetamines, methamphetamine, and opiates at screening or baseline visit
* Participants with a body weight of less than 40 kg
* Consumption of food or drinks containing grapefruit juice, cranberry, pomegranate, star fruit, grapefruit, pomelos, exotic citrus fruits or Seville orange or of alcohol within 72 hours before administration of study treatment.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2018-11-04 (Estimated); Study Completion 2018-11-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) Metabolic Measure of Standard Uptake Value Ratio (SUVR) for Whole Brain, Hippocampal and Dorsolateral Prefrontal Cortices | Baseline (Day -3 to Day -1) to Day 28
  The effects of AGN-242071 on brain metabolic activity or glucose metabolism will be determined using the FDG-PET scan by reporting results as SUVR.
Percentage of Participants with Treatment-Emergent Adverse Events (TEAE) | Day 1 to Day 35
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE that occurs during the treatment period will be considered a TEAE if it was not present before the first dose or if it was present but increased in severity during the treatment period.
Percentage of Participants with Changes from Baseline in Clinically Significant Clinical Laboratory Values | Baseline (Day -3 to Day -1) to Day 35
  Clinical laboratory safety tests include Chemistry, Hematology and Urinalysis.
Percentage of Participants with Changes from Baseline in Clinically Significant Vital Signs | Baseline (Day -3 to Day -1) to Day 35
  Vital signs include systolic and diastolic blood pressure, pulse rate, weight, respiration rate, and temperature.
Percentage of Participants with Changes from Baseline in Clinically Significant Electrocardiogram (ECG) Findings | Baseline (Day -3 to Day -1) to Day 35
  A standard 12-lead ECG will be performed.
Percentage of Participants who have Suicidal Ideation or Behaviours as determined by Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline (Day 1) to Day 35
  The C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and suicidal behavior since the last visit.
Clearance of AGN-242071 | Day 1 to Day 28
  Clearance will be determined utilizing a population pharmacokinetic (PK) approach implemented in non-linear mixed effects modeling (NONMEM®) software.
Volume of Distribution of AGN-242071 | Day 1 to Day 28
  Volume of Distribution will be determined utilizing a population PK approach implemented in NONMEM® software.
Cmax: Maximum Plasma concentration for AGN-242071 | Day 28
AUC: Area Under the Curve for AGN-242071 | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Mitalee Tamhane, PhD, Study Director — Allergan
Locations (6):
- United States (6):
  - ATP Clinical Research, Costa Mesa, California
  - Irvine Center for Clinical Research, Irvine, California
  - Synergy Research Centers, Lemon Grove, California
  - Collaborative Neuroscience, Long Beach, California
  - Alliance Research, Long Beach, California
  - Syrentis Clinical Research, Santa Ana, California